CLINICAL TRIAL: NCT00400634
Title: Multicenter, Randomized, Double-Blind, Sham Surgery-Controlled Study of CERE-120 (Adeno-Associated Virus Serotype 2 [AAV2]-Neurturin [NTN]) to Assess the Efficacy and Safety of Bilateral Intraputaminal (IPu) Delivery in Subjects With Idiopathic Parkinson's Disease
Brief Title: Double-Blind, Multicenter, Sham Surgery Controlled Study of CERE-120 in Subjects With Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Collaborators: Ceregene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CERE-120-02
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2019-08

CONDITIONS: Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intracerebral administration of CERE-120
  Interventions: Drug: CERE-120 (Adeno-Associated Virus Serotype 2 [AAV2]-Neurturin [NTN])
- 2 (Sham Comparator): Sham Neurosurgery
  Interventions: Procedure: Sham Surgery

INTERVENTIONS:
Drug: CERE-120 (Adeno-Associated Virus Serotype 2 [AAV2]-Neurturin [NTN]) — CERE-120 5.4 x 10^11 vg
  Arms: 1
Procedure: Sham Surgery — Bilateral partial thickness burr holes placed, no intraparenchymal injections
  Arms: 2

SUMMARY:
The purpose of this double blind study is to determine whether CERE-120 (adeno-associated virus serotype 2 [AAV2]-neurturin [NTN]) is effective and safe in the treatment of patients with idiopathic Parkinson's Disease. CERE-120 is administered via bilateral stereotactic injections targeting the putaminal region of the brain. The design of this study involves approximately 34 patients receiving CERE-120 treatment via stereotactic surgery and approximately 17 patients receiving sham stereotactic surgery (no CERE-120 administered).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bilateral, idiopathic Parkinson's Disease (PD) based on UK Brain Bank criteria with motor complications despite adequate oral antiparkinsonian therapy.
* At least 5 years disease duration, relative to the anticipated date of surgery, since diagnosis of PD.
* Males or nonpregnant females 35-75 years of age, inclusive.
* A UPDRS motor scale score of 30 or greater in the practically defined off condition during the 30-day eligibility evaluation period.
* Stable doses of antiparkinsonian medications and parkinsonian features for the 60-day period preceding the surgical procedure.
* No conditions that would render the subject unsuitable for surgery, or that would interfere with any of the assessments of efficacy or safety in this trial.
* Subject's informed consent prior to the performance of any study-specific procedures.

Exclusion Criteria:

* Subjects with atypical or secondary parkinsonism.
* Any subject, in the judgment of the investigator, for whom participation in the study would pose a safety risk including, but not limited to, a history of any clinically significant medical, psychiatric, or laboratory abnormality.
* History of treatment of PD by any procedure involving intracranial surgery or implantation of a device.
* MRI of the brain within 12 months before the surgical procedure that indicates the presence of an abnormality that may interfere with the assessments of safety or efficacy or would, in the judgment of the investigator, represent a surgical risk to the subject.
* Any disorder that precludes a surgical procedure (e.g., signs of sepsis or inadequately treated infection) or alters wound healing.
* Receipt of antiplatelet agents for at least 10 days prior to the surgical procedure.
* A score of less than or equal to 27 on the Folstein Mini-Mental examination performed during the eligibility evaluation period or clinical evidence of cognitive impairment that would affect the subject's ability to sign the informed consent or perform any of the protocol required assessments.
* Chemotherapy, cytotoxic therapy, or immunotherapy within 6 weeks prior to the surgical procedure.
* Vaccinations within 30 days prior to the surgical procedure.
* History, within 2 years before the surgical procedure, of drug or alcohol abuse.
* Treatment with neuroleptics within 1 year before the surgical procedure.
* Any medical disability (e.g., severe degenerative arthritis, compromised nutritional state, peripheral neuropathy) that would interfere with the assessment of efficacy and safety in this trial or would compromise the ability of the subject to undergo study procedures (e.g., MRI, PET), or give informed consent.
* History of prior gene transfer therapy.
* Treatment with an investigational agent within 60 days before the surgical procedure.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joao Siffert, M.D., Study Director — Ceregene
Locations (9):
- United States (9):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Rush University Medical Center, Chicago, Illinois
  - Mount Sinai School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Result] Marks WJ Jr, Bartus RT, Siffert J, Davis CS, Lozano A, Boulis N, Vitek J, Stacy M, Turner D, Verhagen L, Bakay R, Watts R, Guthrie B, Jankovic J, Simpson R, Tagliati M, Alterman R, Stern M, Baltuch G, Starr PA, Larson PS, Ostrem JL, Nutt J, Kieburtz K, Kordower JH, Olanow CW. Gene delivery of AAV2-neurturin for Parkinson's disease: a double-blind, randomised, controlled trial. Lancet Neurol. 2010 Dec;9(12):1164-1172. doi: 10.1016/S1474-4422(10)70254-4. Epub 2010 Oct 20. PMID 20970382

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 58 subjects were recruited over a 10.5 month period at 11 centers in the US
Groups:
- CERE-120 Treatment Group: Subjects who were randomized to receive bilateral intraputaminal administration of CERE-120 (5.4 x 10^11 vg)
- Sham Surgery Control Group: Subjects who were randomized to undergo sham surgery (partial burr holes)
Period: Overall Study
Arm/Group | CERE-120 Treatment Group | Sham Surgery Control Group
Started | 38 | 20
Completed | 34 | 19
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CERE-120 Treatment Group | Sham Surgery Control Group | Total
Number analyzed (Participants) | 38 | 20 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (7.56) | 57.3 (8.3) | 59.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 28 | 15 | 43
Region of Enrollment [Number; unit: participants]
  United States | 38 | 20 | 58

OUTCOME MEASURES:

1. Primary Outcome: UPDRS Part III OFF
Description: The UPDRS (Unified Parkinson's Disease Rating Scale) is a clinical rating scale that assesses the symptomatic burden of Parkinson's Disease. The scale has four main sections, and each item is scored from a 0 to a 4 (higher number is more severe manifestation). Part III is a subsection devoted to motor function, has 14 questions, resulting in a score range of 0 (unaffected) to 56 (severely affected). The scale is administered by a trained clinician, and patients were assessed in a practically defined "off" condition, 12 hours or more after the last administration of medication.
Time Frame: Change from Baseline to 12 Month Visit
Population: Subjects who completed the end-of-study visit at month 12 and had no important protocol deviations that potentially could have affected the efficacy assessment of the study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CERE-120 Treatment Group | Sham Surgery Control Group
Number analyzed (Participants) | 34 | 19
units on a scale | -7.21 [-10.34 to -4.09] | -6.91 [-11.16 to -2.66]

2. Other Pre Specified Outcome: UPDRS Part III OFF
Description: as for outcome 1
Time Frame: Change from Baseline to 18 Month Visit
Population: Subjects who completed the 12-month double-blind posttreatment period of the study continued to undergo double-blind assessments every 3 months until the last subject had completed the end-of-study visit at month 12. The LOCF method was used to impute data at month 18 for the subjects who had blinded data through month 15.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CERE-120 Treatment Group | Sham Surgery Control Group
Number analyzed (Participants) | 19 | 11
units on a scale | -11.96 (7.068) | -4.34 (2.479)

ADVERSE EVENTS:
Time Frame: 23 months
Arm/Group | CERE-120 Treatment Group | Sham Surgery Control Group
Serious Adverse Events (participants affected / at risk) | 13/38 | 4/20
Other Adverse Events (participants affected / at risk) | 38/38 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CERE-120 Treatment Group (N=38) | Sham Surgery Control Group (N=20)
Death (Vascular disorders) | 2 (2) | 0 (0) — Neither death was considered related to CERE-120
spinal compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not considered related to CERE-120
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Considered not related to CERE-120
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Considered not related to CERE-120
Urinary Retention (Renal and urinary disorders) | 2 (2) | 0 (0) — Considered not related to CERE-120
Lumbar Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Considered not related to CERE-120
Cerebral Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) — Considered not related to CERE-120, Related to surgical procedure
Gait Disturbance (Nervous system disorders) | 1 (1) | 0 (0) — Not considered related to CERE-120
Nerve Root Compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Considered not related to CERE-120
Device Failure (Surgical and medical procedures) | 1 (1) | 0 (0) — Considered not related to CERE-120
Esophageal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Considered not related to CERE-120
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fall (Nervous system disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CERE-120 Treatment Group (N=38) | Sham Surgery Control Group (N=20)
Headache (Nervous system disorders) | 28 | 10
Dyskinesia (Nervous system disorders) | 9 | 6
Parkinson's Disease (Nervous system disorders) | 8 | 4
Dizziness (Nervous system disorders) | 4 | 4
Hypoaesthesia (Nervous system disorders) | 1 | 4
Tremor (Nervous system disorders) | 2 | 2
Freezing Phenomena (Nervous system disorders) | 2 | 1
Balance Disorder (Nervous system disorders) | 2 | 0
Brain Edema (Nervous system disorders) | 2 | 0
Cognitive Disorder (Nervous system disorders) | 2 | 0
Post Procedural Pain (Injury, poisoning and procedural complications) | 11 | 7
Headache Postoperative (Injury, poisoning and procedural complications) | 5 | 5
Incision Site Complication (Injury, poisoning and procedural complications) | 6 | 2
Fall (Injury, poisoning and procedural complications) | 4 | 2
Procedural Hypotension (Injury, poisoning and procedural complications) | 3 | 0
Nausea (Gastrointestinal disorders) | 13 | 6
Constipation (Gastrointestinal disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 0
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 8 | 2
Depression (Psychiatric disorders) | 4 | 3
Anxiety (Psychiatric disorders) | 2 | 4
Confusional State (Psychiatric disorders) | 1 | 2
Hallucinations (Psychiatric disorders) | 3 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 2
Bronchitis (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 3 | 0
Gastroenteritis (Infections and infestations) | 0 | 2
Fatigue (General disorders) | 3 | 1
Face Edema (General disorders) | 2 | 1
Gait Disturbance (General disorders) | 2 | 1
Edema (General disorders) | 2 | 0
Edema Peripheral (General disorders) | 2 | 0
Micturation Urgency (Renal and urinary disorders) | 4 | 1
Hematuria (Renal and urinary disorders) | 3 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 1
Urinary Incontinence (Renal and urinary disorders) | 3 | 0
Urinary Retention (Renal and urinary disorders) | 3 | 0
Renal Failure (Renal and urinary disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 0
Periorbital Edema (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 0
Blood Testosterone Decreased (Investigations) | 2 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sleep Apnea Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypertension (Vascular disorders) | 3 | 2
Hypotension (Vascular disorders) | 2 | 1
Vision Blurred (Eye disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days